CLINICAL TRIAL: NCT04090580
Title: Impact on Glycemic Variability in Newly Onset T2DM Patients Initiating Dapagliflozin Plus Metformin Versus Metformin Alone: A Randomized Open Label Clinical Study. The MAGNNIFY Trial.
Brief Title: Impact on Glycemic Variability in Newly Onset T2DM Patients Initiating Dapagliflozin Plus Metformin Versus Metformin Alone
Acronym: MAGNNIFY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Miguel Ángel Gómez Sámano, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3089
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: dapagliflozin; glycemic variability; MAGE; DIABETES MELLITUS
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Evaluation of efficacy between Dapagliflozin with Metformin (Intervention) vs Metformin alone (Standard of care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAPAGLIFLOZIN 10 mg/day + METFORMIN 2000 mg/day for 12 weeks (Experimental): Subjects enrolled will be randomized 1:1 to receive a daily dosage of 10 mg dapagliflozin and 2000 mg metformin for 12 weeks
  Interventions: Diagnostic Test: Continuous glucose monitoring
- METFORMIN 2000 mg/day for 12 weeks (Active Comparator): Subjects enrolled will be randomized 1:1 to receive a daily dosage of 2000 mg Metformin for 12 weeks
  Interventions: Diagnostic Test: Continuous glucose monitoring

INTERVENTIONS:
Diagnostic Test: Continuous glucose monitoring — Subjects enrolled will be randomized 1:1 to either receive a daily dosage of dapagliflozin 10 mg and 2000 mg metformin for 12 weeks or 2000 mg metformin. Patients who do not tolerate metformin at 2000mg dose will be downtitrated to 1500 mg daily. In case patients do not tolerate 1500 mg daily, they will be excluded.
  Both groups will be monitored for 7 days using either iPro™ CGM system (Medtronic, Northridge, CA) or Dexcom G6 CGM (Dexcom Inc, San Diego, CA). Basal continuous glucose monitoring will start at week 1 (first visit), and removed at day 7 and final continuous glucose monitoring will start at week 11 and removed 7 days after (final visit).

SUMMARY:
This study will compare the effect of Dapagliflozin added to Metformin vs Metformin alone on blood sugar fluctuations of adults with a recent diagnosis of Type 2 Diabetes (T2D). The duration of the protocol will be 12 weeks. Continuous glucose monitoring will be measured before and at the end of the intervention. The questions this protocol will answer include:

* Is there a difference in blood sugar fluctuations when Dapagliflozin is added to Metformin compared with Metformin alone in adults with type 2 Diabetes?
* Does Dapagliflozin added to Metformin improve blood glucose control in patients with type 2 Diabetes?

DETAILED DESCRIPTION:
This is an open-label randomized clinical trial aimed to compare the effect of Dapagliflozin added to Metformin vs Metformin alone on glycemic variability of adults with a recent diagnosis of type 2 Diabetes. The central hypothesis is that the addition of Dapagliflozin will lead to a statistically significant improvement in GV parameters compared to Metformin alone. A total of 88 adults aged 18-70 years with T2DM and HbA1c between 7.5% and 12% while on a stable dose of Metformin 2000 mg/day will be enrolled. Participants will be randomized in a 1:1 ratio to one of two treatment arms for a duration of 12 weeks. The primary objective is to compare the change from baseline to end-of-treatment in key glycemic variability indices derived from continuous glucose monitoring (CGM) (Mean Amplitude Glucose Excursions -MAGE, Time in Range), changes in HbA1c, fasting blood glucose, lipid profile, BMI, blood pressure, among others.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18-77 years-old
* Both Male and female
* Hba1c ≥ 7.5 % and ≤12%
* BMI > 25 and <45 kg/m2
* Type 2 diabetes diagnosis, drug-naive

Exclusion Criteria:

* Hba1c > 12%
* Creatinine clearance CKD-EPI: < 60 mL/min
* LADA or Type 1 diabetes
* Gestational diabetes
* Clinically significant disease like: hepatic, hematological, oncological, psychiatric or rheumatic disease.
* Symptoms of marked uncontrolled diabetes: (marked poliuria or polidipsia + 10% weight loss prior the last 3 months enrollement)
* Known hypersensitivity to dapagliflozin or any of the excipients of the product
* eGFR persistently <45 mL/min/1.73 m2
* Unstable or rapidly progressing renal disease
* Patients with severe hepatic impairment (Child-Pugh class C)
* Any major CV event/Vascular Disease within 3 months prior to signing the consent at enrollment, as assessed by the investigator
* For women only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Gomez Samano, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán ''INCMNSZ'', Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Participants were identified with name and last names initials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment began in October 2019 and was interrupted due to the SARS-COV-2 pandemic in March 2020. Nevertheless, patients who were already enrolled were followed up. Recruitment was normally restarted in March 2021; one of the inclusion criteria was adjusted, allowing HbA1c <13.0%, prior limit <12.0%. The last patient was recruited on December 6th, 2021.The complete study was concluded on March 2021.
Pre-assignment Details: Treatment: subjects who met the pre-randomization period and tolerated treatment were randomized 1:1 to receive either DAPA 10 mg/day + MET 2000 mg/day or MET 2000 mg/day for 12 weeks.
  Of the total of 264 patients surveyed, a sample of 88 met the inclusion criteria and none of the exclusion criteria randomization DAPA+MET n=42 and MET n= 46
Groups:
- DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks: Subjects enrolled will be randomized 1:1 to either receive a daily dosage of 10 mg dapagliflozin and 2000 mg metformin for 12 weeks
  Continuous glucose monitoring: Subjects enrolled will be randomized 1:1 to either receive a daily dosage of dapagliflozin 10 mg and 2000 mg metformin for 12 weeks (n=18) or 2000 mg metformin (n=18). Patients who do not tolerate metformin at 2000mg dose will be downtitrated to 1500 mg daily. In case patients do not tolerate 1500 mg daily, they will be excluded.
  Both groups will be monitored for 7 days using either iPro™ CGM system (Medtronic, Northridge, CA) or Dexcom G6 CGM (Dexcom Inc, San Diego, CA). Basal continuous glucose monitoring will start at week 1 (first visit), and removed at day 7 and final continuous glucose monitoring will start at week 11 and removed 7 days after (final visit).
- METFORMIN 2000 mg/Day for 12 Weeks: Subjects enrolled will be randomized 1:1 to either receive a daily dosage of 2000 mg metformin for 12 weeks
  Continuous glucose monitoring: Subjects enrolled will be randomized 1:1 to either receive a daily dosage of dapagliflozin 10 mg and 2000 mg metformin for 12 weeks (n=18) or 2000 mg metformin (n=18). Patients who do not tolerate metformin at 2000mg dose will be downtitrated to 1500 mg daily. In case patients do not tolerate 1500 mg daily, they will be excluded.
  Both groups will be monitored for 7 days using either iPro™ CGM system (Medtronic, Northridge, CA) or Dexcom G6 CGM (Dexcom Inc, San Diego, CA). Basal continuous glucose monitoring will start at week 1 (first visit), and removed at day 7 and final continuous glucose monitoring will start at week 11 and removed 7 days after (final visit).
Period: Overall Study
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Started | 42 | 46
Completed | 41 | 39
Not Completed | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks | Total
Number analyzed (Participants) | 42 | 46 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 46 | 88
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (8.6) | 50.9 (11.8) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 20 | 23 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 46 | 88
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 42 | 46 | 88
MAGE mmol/L [Mean (Standard Deviation); unit: mmol/L] | 4.3 (1.2) | 4.1 (1.5) | 4.2 (1.3)
weight kg [Mean (Standard Deviation); unit: kg] | 81.3 (19.1) | 80.0 (13.9) | 80.5 (16)
HbA1c% [Mean (Standard Deviation); unit: %] | 9.2 (1.6) | 9.4 (1.3) | 9.3 (1.4)
insulin µU/mL [Mean (Standard Deviation); unit: µU/mL] | 12.2 (13.3) | 10.9 (6.6) | 11 (9)
triglycerides mg/dL [Mean (Inter-Quartile Range); unit: mg/dL] | 193 [135.2 to 271.2] | 185.5 [135.2 to 240] | 190 [135 to 265]
uric acid mg/dL [Mean (Standard Deviation); unit: mg/dL] | 5.7 (1.3) | 5.4 (1.4) | 5.5 (1.3)
SBP mm/Hg [Mean (Standard Deviation); unit: mm/Hg] | 136.1 (21.8) | 130.8 (16.6) | 133 (18)
TIR %target 70-180 mg/dL [Mean (Inter-Quartile Range); unit: %] | 55.5 [12.6 to 80.6] | 82.7 [26.1 to 95.1] | 69.1 [18 to 87]

OUTCOME MEASURES:

1. Primary Outcome: ΔHbA1c
Description: Difference between serum HbA1c before treatment (W0) and at the end of intervention (W12) expressed in percentage.
Time Frame: 12 weeks
Population: In the intention to treat analysis (ITT), early T2DM treatment with DAPA+MET (n=42) resulted in significant improvements in several health indicators compared to patients in the MET group (n=46). Results are presented as Δ, which represents the change between W0 and W12 values
Measure: Mean (Inter-Quartile Range); unit: percentage of HbA1c
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Number analyzed (Participants) | 42 | 46
percentage of HbA1c | -1.8 [-3 to -0.5] | -1.6 [-2.9 to 0]

2. Primary Outcome: ΔMAGE
Description: ● Calculation of Mean Amplitude of Glucose Excursion (MAGE):
  * In the first step, all local maximum/minimum values are determined.
  * The next step is an evaluation of maximum/minimum pairs against the standard deviation (SD).
  * If the difference from minimum to maximum is greater than the SD, this variation from the mean measurement is retained.
  * If the local maximum/minimum is less than 1 SD, it is excluded from further calculations.
  * These channels are retained and summed to achieve the MAGE
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: mmol/dL
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Number analyzed (Participants) | 42 | 46
mmol/dL | -0.8 [-1.6 to 0.0] | 0.0 [-1.1 to 0.6]

3. Primary Outcome: Δweight
Description: The difference between weight before the treatment period (W0) and the end of the intervention is calculated and expressed as delta for results interpretation.
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: kg
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Number analyzed (Participants) | 42 | 46
kg | -2.7 [-4.40 to -1.40] | -0.7 [-2.6 to 0.55]

4. Primary Outcome: ΔTIR %Target 70-180 mg/dL
Description: Time in range is defined as the percentage of time that the patient's blood glucose is between 70-180 mg/dL.
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: percentage of time
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Number analyzed (Participants) | 42 | 46
percentage of time | 31.5 [3.6 to 72.3] | 0.4 [-8.5 to 39.2]

5. Primary Outcome: Δinsulin
Description: Delta insulin is defined as the difference in insulin plasma concentration before treatment (W0) and at the end of the intervention (W12).
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: uU/mL
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Number analyzed (Participants) | 42 | 46
uU/mL | -2.5 [-4.5 to -0.6] | 0.4 [-1.0 to 4.5]

6. Primary Outcome: Δsystolic Blood Pressure
Description: It is defined as the difference in systolic blood pressure before treatment (W0) and after the end of intervention (W12)
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: mm/Hg
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Number analyzed (Participants) | 42 | 46
mm/Hg | -2.0 [-15.0 to 5.0] | 0.0 [-13.0 to 15.0]

7. Primary Outcome: ΔTriglycerides mg/dL
Description: It is defined as the difference in triglycerides plasma concentration before and at the end of intervention (W12-W0)
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Number analyzed (Participants) | 42 | 46
mg/dL | -50.5 [-103.0 to 2.2] | -21.5 [-680 to 23.0]

8. Secondary Outcome: ΔUric Acid
Description: It is defined as the difference in plasma uric acid concentration before and at the end of intervention (W12-W0)
Time Frame: 12 weeks
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
Number analyzed (Participants) | 42 | 46
mg/dL | -0.4 [-1.4 to 0.0] | 0.0 [-0.2 to 0.6]

ADVERSE EVENTS:
Time Frame: From the start of the intervention until the end of treatment, 12 weeks.
Description: Number of participants at risk for Serious Adverse Events: 88 participants Number of participants at risk for All-Cause Mortality: 88 participants Number of participants at risk for Other Adverse Events: 88 participants
Arm/Group | DAPAGLIFLOZIN 10 mg/Day + METFORMIN 2000 mg/Day for 12 Weeks | METFORMIN 2000 mg/Day for 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/46
Other Adverse Events (participants affected / at risk) | 0/42 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04090580/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04090580/SAP_003.pdf
  • Informed Consent Form (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT04090580/ICF_004.pdf